CLINICAL TRIAL: NCT07220252
Title: Ublituximab in Pediatric Participants With Relapsing Forms of Multiple Sclerosis (RMS)
Brief Title: Study to Assess Effects of Ublituximab in Pediatric Participants With Relapsing Forms of Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG1101-RMS-PED304; 2025-522257-19-00 (Other: EU CT Number)
Record Dates: First submitted 2025-10-22; First posted 2025-10-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ublituximab; Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Ublituximab (Experimental): New Regimen
  Interventions: Drug: Ublituximab
- Part B: Ublituximab (Experimental): New Regimen
  Interventions: Drug: Ublituximab
- Part B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B: Fingolimod (Experimental)
  Interventions: Drug: Fingolimod
- Part B: IV Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part C: OLE (Experimental)
  Interventions: Drug: Ublituximab

INTERVENTIONS:
Drug: Ublituximab — Administered as an intravenous (IV) infusion.
  Other Names: TG-1101; BRIUMVI
  Arms: Part A: Ublituximab; Part B: Ublituximab; Part C: OLE
Drug: Placebo — Oral capsule.
  Arms: Part B: Placebo
Drug: Placebo — IV infusion.
  Arms: Part B: IV Placebo
Drug: Fingolimod — Oral capsule.
  Arms: Part B: Fingolimod

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of ublituximab in participants ages 10 to less than (<)18 years and body weight greater than or equal to (≥)25 kilograms (kg) to less than or equal to (≤)40 kg with RMS (Part A) and to evaluate the non-inferiority of ublituximab compared with fingolimod in pediatric RMS participants with body weight ≥ 25 kg (Part B). The study will further evaluate long-term safety and efficacy of ublituximab in RMS in pediatric participants during its extension period (Part C).

ELIGIBILITY:
Inclusion Criteria for Part A and Part B:

1. Diagnosis of RMS.
2. EDSS at screening: 0-5.5, inclusive.
3. Neurologic stability for ≥ 30 days prior to screening, and between screening and Week 1 Day 1 (W1D1).

Inclusion Criteria for Part C:

1. Participants must have completed Part A (Week 24 visit) or Part B (Week 96 visit) to be eligible for Part C.

Exclusion Criteria for Part A and B:

1. Known presence or suspicion of other neurologic disorders that may mimic MS.
2. Prior treatments:

   1. Systemic corticosteroids (>0.1 milligrams/kilogram/day [mg/kg/day], or >5 milligrams/day [mg/day] of prednisone equivalent) or adrenocorticotropic hormone (ACTH) within 30 days prior to the screening MRI scan (note: Topical, ophthalmic, or inhaled corticosteroids are permitted).
   2. High dose intravenous immunoglobulin (IVIG) or subcutaneous IG (SCIG) within 2 months prior to W1D1.
   3. Treatment with anti-CD20 or other B cell directed treatment at any time.
   4. Treatment with alemtuzumab, cladribine, cyclophosphamide, mitoxantrone at any time.

Additional Exclusion Criteria for Part B Only (Relevant to Fingolimod Treatment):

1. Treatment with fingolimod or other sphingosine-1 phosphate-1 (S1P1) modulators at any time.
2. The following antiarrhythmic drugs at Screening: Class Ia anti-arrhythmics.

Exclusion Criteria for Part C:

1. If the absolute lymphocyte count (ALC) is outside the specified range the participant will not be eligible to receive ublituximab in Part C.

Note: Other protocol-specified inclusion/exclusion criteria may apply

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Area Under the Curve From Week 0 to 24 (AUC0-W24) of Ublituximab | Predose and multiple timepoints up to Week 24
Part A: Maximum Observed Concentration (Cmax) of Ublituximab | Day 1 and Day 15
Part A: Participant B Cell Counts | Up to Week 24
Part B: Annualized Relapse Rate (ARR) | Up to 96 weeks
Part C: Annualized Relapse Rate (ARR) | Up to 168 weeks

SECONDARY OUTCOMES:
Part A, B and C: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Part A: Up to Week 24; Part B: Up to 96 weeks; Part C: Up to 168 weeks
Part A, B and C: Number of Participants With Change in Columbia-Suicide Severity Rating Scale (C-SSRS ) | Part A: Up to Week 24; Part B: Up to 96 weeks; Part C: Up to 168 weeks
Part A: Serum Concentrations of Ublituximab | Up to Week 24
Part A and B: Percentage of Participants with Treatment-emergent Anti-drug Antibodies (ADAs) to Ublituximab | Part A: Up to Week 24; Part B: Up to 96 weeks
Part A and B: Number of Gadolinium Enhancing (Gd-enhancing) T1 Lesions per Magnetic Resonance Imaging (MRI) Scan | Part A: Up to Week 24; Part B: Up to 96 weeks
Part A and B: Number of New and/or enlarging T2 Hyperintense Lesions (NELs) per MRI Scan | Part A: Up to Week 24; Part B: Up to 96 weeks
Past A: Annualized Relapse Rate | Up to Week 24
Part A and C: Change From Baseline in Expanded Disability Status Scale (EDSS) Score | Part A: Baseline, up to Week 24; Part C: Baseline, up to 168 weeks
Part B: Pharmacokinetics (PK) Serum Concentration of Ublituximab | Up to Week 96
Part B: Percentage of Participants with CD19+ B cell counts ≤10 cells/uL | Up to 96 weeks
Part B: Annualized Relapse Rate ARR | Up to Week 96
Part C: Time to Confirmed Disability Progression (CDP) | Up to Week 24
Part C: Time to Confirmed Disability Improvement (CDI) | Up to Week 24

IPD SHARING:
Plan to Share IPD: No